CLINICAL TRIAL: NCT06917118
Title: Multimodal Pain Management After Wide Awake Local Anesthesia No Tourniquet Orthopedic Hand Surgery: A Randomized Control Trial
Acronym: WALANT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Daniel Deliz, Dr. Christian A. Foy, University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2501339638
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Pain Management
Keywords: WALANT; Multimodal analgesia; Nonopioid pain management; VAS pain scores
MeSH Terms: conditions — Agnosia | interventions — Oxycodone; Acetaminophen; Naproxen; Tablets

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Postoperative opioid analgesia (Active Comparator): 10 pills of 5mg oxycodone Q4hrs as needed
  Interventions: Drug: Oxycodone 5mg taken first
- Postoperative Opioid-sparing Multimodal analgesia (Experimental): 30 pills of 500mg acetaminophen Q4hrs and 30 pills of 500mg naproxen Q4hrs. Will also receive 5 tablets of 5mg oxycodone to take Q4hrs as needed for breakthrough pain
  Interventions: Drug: Acetaminophen; Drug: Naproxen Tablets, 500 mg; Drug: OxyCODONE 5 mg Oral Tablet

INTERVENTIONS:
Drug: Oxycodone 5mg taken first — 10 pills of 5mg oxycodone Q4hrs as needed
  Arms: Standard Postoperative opioid analgesia
Drug: Acetaminophen — 30 pills of 500mg acetaminophen Q4hrs
  Arms: Postoperative Opioid-sparing Multimodal analgesia
Drug: Naproxen Tablets, 500 mg — 30 pills of 500mg naproxen Q4hrs
  Arms: Postoperative Opioid-sparing Multimodal analgesia
Drug: OxyCODONE 5 mg Oral Tablet — Only used for breakthrough pain
  Arms: Postoperative Opioid-sparing Multimodal analgesia

SUMMARY:
The main objective of the study is to measure the efficacy of a multimodal postoperative pain regimen consisting of oral acetaminophen and naproxen compared to a traditional opioid-only pain regimen following elective wide awake local anesthesia no tourniquet (WALANT) hand surgery in a Hispanic population. The study is a randomized control trial comparing the clinical outcomes of patients undergoing elective WALANT hand surgery performed by a board-certified, fellowship-trained orthopedic hand surgeon (Dr. Christian A. Foy).

The study groups are:

* Control group: standard pain control with opioids
* Experimental group: multimodal non-opioid pain control

Study Outcomes are:

* VAS pain scores (7 days),
* Total opioid usage
* Patient satisfaction
* Adverse events

We hypothesize that patients receiving multimodal pain regimens will report lower opioid use, lower pain scores, and greater satisfaction than patients receiving traditional opioid-only pain management.

DETAILED DESCRIPTION:
The main objective of the study is to measure the efficacy of a multimodal postoperative pain regimen consisting of oral acetaminophen and naproxen compared to a traditional opioid-only pain regimen following elective wide awake local anesthesia no tourniquet (WALANT) hand surgery in a Hispanic population. The study is a single-blind, single-center randomized control trial comparing the clinical outcomes of patients undergoing elective WALANT hand surgery performed by a board-certified, fellowship-trained orthopedic hand surgeon (Dr. Christian A. Foy). Patients will be consecutively recruited at the center and randomized in a 1:1 ratio into the control and experimental groups. The control group will receive the standard of care for postoperative pain: 10 pills of 5mg oxycodone Q4hrs as needed. The experimental group will receive 30 pills of 500mg acetaminophen Q4hrs and 30 pills of 500mg naproxen Q4hrs until pain resolves or treatment is completed. The experimental group will also receive 5 tablets of 5mg oxycodone to take Q4hrs as needed for breakthrough pain. Postoperatively, daily pain Visual Analog Scale (VAS) scores, total opioid usage, patient satisfaction, and adverse events will be recorded. We hypothesize that patients receiving multimodal pain regimens will report lower opioid use, lower pain scores, and greater satisfaction than patients receiving traditional opioid-only pain management.

ELIGIBILITY:
Inclusion Criteria:

* Patients 21-70 years of age undergoing outpatient hand surgery
* Patients undergoing surgery with WALANT technique
* Patients who provide written informed consent

Exclusion Criteria:

* Patients aged 20 and younger, or 71 and older
* Patient with chronic pain requiring opioid use
* Pregnant patients
* Patients who do not self-identify as Hispanic
* Patients with known allergy to the medication
* Patients with contraindications for the prescribed medications

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
VAS Pain Scores | From enrollment to the end of treatment at 7 days
  VAS pain scores will be assessed using a patient- completed VAS pain questionnaire until 7 days post-op. Patients will take the questionnaire home and report pain scores in the morning and in the afternoon every day for a week.
Patient Satisfaction | From enrollment to the end of treatment at 7 days
  Patient satisfaction will be assessed using the Patient Satisfaction Questionnaire Short Form (PSQ-18)
Total Opioid Usage | From enrollment to the end of treatment at 7 days
  Will be reported in as morphine milligram equivalents (MMEs)

SECONDARY OUTCOMES:
Breakthrough Pain | From enrollment to the end of treatment at 7 days
  Breakthrough pain will be reported as a binary outcome (Y/N)
Length of Treatment | From enrollment to the end of treatment at 7 days
  Patients will be asked to report the number of days in which they used the provided pain control treatment
Indication for WALANT surgery | From enrollment to the end of treatment at 7 days
  We will report the indication for treatment for each patient to include in the final analysis

CONTACTS AND LOCATIONS:
Overall Officials: Christian A. Foy, MD, Principal Investigator — University of Puerto Rico Medical Sciences Campus
Locations (1):
- Oncological Hospital, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will only be used internally by the study PI and primary investigators.

REFERENCES:
- [Background] Abdullah S, Ahmad AA, Lalonde D. Wide Awake Local Anesthesia No Tourniquet Forearm Triple Tendon Transfer in Radial Nerve Palsy. Plast Reconstr Surg Glob Open. 2020 Aug 11;8(8):e3023. doi: 10.1097/GOX.0000000000003023. eCollection 2020 Aug. PMID 32983779
- [Background] Burn MB, Shapiro LM, Eppler SL, Behal R, Kamal RN. Clinical Care Redesign to Improve Value for Trigger Finger Release: A Before-and-After Quality Improvement Study. Hand (N Y). 2021 Sep;16(5):624-631. doi: 10.1177/1558944719884661. Epub 2019 Nov 5. PMID 31690136
- [Background] Lalonde D, Bell M, Benoit P, Sparkes G, Denkler K, Chang P. A multicenter prospective study of 3,110 consecutive cases of elective epinephrine use in the fingers and hand: the Dalhousie Project clinical phase. J Hand Surg Am. 2005 Sep;30(5):1061-7. doi: 10.1016/j.jhsa.2005.05.006. PMID 16182068
- [Background] Chowdhry S, Seidenstricker L, Cooney DS, Hazani R, Wilhelmi BJ. Do not use epinephrine in digital blocks: myth or truth? Part II. A retrospective review of 1111 cases. Plast Reconstr Surg. 2010 Dec;126(6):2031-2034. doi: 10.1097/PRS.0b013e3181f44486. PMID 20697319
- [Background] Sawhney A, Thacoor A, Nagra R, Geoghegan L, Akhavani M. Wide Awake Local Anesthetic No Tourniquet in Hand and Wrist Surgery: Current Concepts, Indications, and Considerations. Plast Reconstr Surg Glob Open. 2024 Jan 22;12(1):e5526. doi: 10.1097/GOX.0000000000005526. eCollection 2024 Jan. PMID 38260757
- [Background] Deutsch CJ, Jones K, Dassayanake S, Milroy C. Concern about ischaemia drives a persistent and generation-spanning aversion to adrenaline in digital anaesthesia. JPRAS Open. 2021 Jan 26;28:61-63. doi: 10.1016/j.jpra.2021.01.006. eCollection 2021 Jun. No abstract available. PMID 33732855
- [Background] Fillingham YA, Hannon CP, Erens GA; AAHKS Anesthesia & Analgesia Clinical Practice Guideline Workgroup; Hamilton WG, Della Valle CJ. Acetaminophen in Total Joint Arthroplasty: The Clinical Practice Guidelines of the American Association of Hip and Knee Surgeons, American Society of Regional Anesthesia and Pain Medicine, American Academy of Orthopaedic Surgeons, Hip Society, and Knee Society. J Arthroplasty. 2020 Oct;35(10):2697-2699. doi: 10.1016/j.arth.2020.05.030. Epub 2020 May 26. No abstract available. PMID 32571591
- [Background] Padilla JA, Gabor JA, Schwarzkopf R, Davidovitch RI. A Novel Opioid-Sparing Pain Management Protocol Following Total Hip Arthroplasty: Effects on Opioid Consumption, Pain Severity, and Patient-Reported Outcomes. J Arthroplasty. 2019 Nov;34(11):2669-2675. doi: 10.1016/j.arth.2019.06.038. Epub 2019 Jun 26. PMID 31311667
- [Background] Gimbel JS, Brugger A, Zhao W, Verburg KM, Geis GS. Efficacy and tolerability of celecoxib versus hydrocodone/acetaminophen in the treatment of pain after ambulatory orthopedic surgery in adults. Clin Ther. 2001 Feb;23(2):228-41. doi: 10.1016/s0149-2918(01)80005-9. PMID 11293556
- [Background] Thompson KA, Klein D, Alaia MJ, Strauss EJ, Jazrawi LM, Campbell KA. Opioid Use Is Reduced in Patients Treated with NSAIDs After Arthroscopic Bankart Repair: A Randomized Controlled Study. Arthrosc Sports Med Rehabil. 2020 Dec 27;3(1):e15-e22. doi: 10.1016/j.asmr.2020.08.003. eCollection 2021 Feb. PMID 33615243
- [Background] Hess-Arcelay H, Claudio-Marcano A, Torres-Lugo NJ, Deliz-Jimenez D, Acosta-Julbe J, Hernandez G, Deliz-Jimenez D, Monge G, Ramirez N, Lojo-Sojo L. Opioid-Sparing Nonsteroid Anti-inflammatory Drugs Protocol in Patients Undergoing Intramedullary Nailing of Tibial Shaft Fractures: A Randomized Control Trial. J Am Acad Orthop Surg. 2024 Jun 15;32(12):e596-e604. doi: 10.5435/JAAOS-D-23-01014. Epub 2024 Apr 4. PMID 38579315
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Chung F, Ritchie E, Su J. Postoperative pain in ambulatory surgery. Anesth Analg. 1997 Oct;85(4):808-16. doi: 10.1097/00000539-199710000-00017. PMID 9322460
- [Background] Pasero C, McCaffery M. Orthopaedic postoperative pain management. J Perianesth Nurs. 2007 Jun;22(3):160-72; quiz 172-3. doi: 10.1016/j.jopan.2007.02.004. PMID 17543801
- [Background] Trasolini NA, McKnight BM, Dorr LD. The Opioid Crisis and the Orthopedic Surgeon. J Arthroplasty. 2018 Nov;33(11):3379-3382.e1. doi: 10.1016/j.arth.2018.07.002. Epub 2018 Jul 11. PMID 30075877
- [Background] Harris JD. Management of expected and unexpected opioid-related side effects. Clin J Pain. 2008 May;24 Suppl 10:S8-S13. doi: 10.1097/AJP.0b013e31816b58eb. PMID 18418226
- [Background] Huynh MNQ, Yuan M, Gallo L, Olaiya OR, Barkho J, McRae M. Opioid Consumption After Upper Extremity Surgery: A Systematic Review. Hand (N Y). 2024 Sep;19(6):1002-1011. doi: 10.1177/15589447231160211. Epub 2023 Mar 23. PMID 36960481
- [Background] Feinberg AE, Chesney TR, Srikandarajah S, Acuna SA, McLeod RS; Best Practice in Surgery Group. Opioid Use After Discharge in Postoperative Patients: A Systematic Review. Ann Surg. 2018 Jun;267(6):1056-1062. doi: 10.1097/SLA.0000000000002591. PMID 29215370
- [Background] Fader L, Whitaker J, Lopez M, Vivace B, Parra M, Carlson J, Zamora R. Tibia fractures and NSAIDs. Does it make a difference? A multicenter retrospective study. Injury. 2018 Dec;49(12):2290-2294. doi: 10.1016/j.injury.2018.09.024. Epub 2018 Sep 18. PMID 30270011
- [Background] Rodgers J, Cunningham K, Fitzgerald K, Finnerty E. Opioid consumption following outpatient upper extremity surgery. J Hand Surg Am. 2012 Apr;37(4):645-50. doi: 10.1016/j.jhsa.2012.01.035. Epub 2012 Mar 10. PMID 22410178